CLINICAL TRIAL: NCT07259707
Title: A Single-Center, Prospective, Single-Arm Phase II Clinical Study of Consolidation With High-Dose Cytarabine Following Deep Molecular Remission Induced by Gilteritinib Plus VA Regimen in Newly Diagnosed Intermediate-Risk Fit AML Patients With FLT3-ITD Mutation
Brief Title: Gilteritinib Plus VA Followed By Consolidation Chemotherapy in Newly Diagnosed FLT3-ITD+ AML
Acronym: GANCE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Jie Sun, Principle Attending, Associated Professor, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250133C
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; FLT3 Internal Tandem Duplication Positive; Intermediate Risk Acute Myeloid Leukemia; Fit Patients
Keywords: acute myeloid leukemia; FLT3-ITD; Intermediate Risk; Fit; Gilteritinib; Deep molecular remission
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GVA + HDAC Consolidation + Gilteritinib Maintenance (Experimental): This is a single-arm study contains three phases:
  Phase I. Induction Therapy: Gilteritinib + Venetoclax + Azacitidine (GVA Regimen) for 2 cycles Phase II. Consolidation Therapy: Gilteritinib + High-Dose Cytarabine (HDAC) for 3 cycles Phase III. Maintenance Therapy: Gilteritinib monotherapy for up to 3 months
  Interventions: Drug: GVA + HDAC Consolidation & Gilteritinib Maintenance

INTERVENTIONS:
Drug: GVA + HDAC Consolidation & Gilteritinib Maintenance — Phase I. Induction Therapy (2 cycles): Gilteritinib plus 80 mg, orally (po), once daily (qd), continuously from Day 1 of Cycle 1 until the end of Induction.Venetoclax + Azacitidine (VA Regimen): Azacitidine: 75 mg/m², intravenously (iv) or subcutaneously (sc), once daily on Days 1-7 of each 28-day cycle.Venetoclax: Cycle 1: Dose ramp-up: 100 mg po on Day 1, 200 mg po on Day 2, then 400 mg po once daily from Day 3 to Day 28.Subsequent Cycles: 400 mg po once daily on Days 1-28 of each 28-day cycle.
  Phase II. Consolidation Therapy (3 cycles): High-Dose Cytarabine (HiDAC): 3.0 g/m², intravenously (iv), over 3 hours, every 12 hours (q12h) on Days 1, 3, and 5 (total of 6 doses per cycle)；Gilteritinib: Dose increased to 120 mg, orally (po), once daily (qd), from day8 to day21. The interval of each cycle is 30 days.
  Phase III. Maintenance Therapy: Gilteritinib: 120 mg, orally (po), once daily (qd), continuously for up to 3 months.

SUMMARY:
This clinical trial aims to evaluate whether molecular MRD-guided chemotherapy can effectively treat FLT3-ITD mutated AML and potentially replace allogeneic hematopoietic stem cell transplantation. It primarily seeks to answer:

* What is the complete remission rate after initial induction with Gilteritinib, Venetoclax, and Azacitidine?
* What are the survival rates and safety of subsequent high-dose cytarabine consolidation after two cycles of this induction therapy? As a single-arm study, outcomes will be compared against historical data from standard treatments (including transplant) to assess if the new strategy is equally or more effective.

Participants will:

* Undergo three cycles of high-dose cytarabine consolidation after two cycles of induction therapy, contingent upon achieving deep FLT3-ITD molecular remission.
* Start Gilteritinib maintenance therapy after consolidation if FLT3-ITD remains detectable, continuing until deep molecular remission is achieved again.

DETAILED DESCRIPTION:
This single-center, phase II trial evaluates a novel, transplant-sparing strategy for fit patients with newly diagnosed intermediate-risk acute myeloid leukemia (AML) harboring FLT3-ITD mutations. The central hypothesis is that achieving deep molecular remission-as measured by a highly sensitive assay termed "DeepScan" (Levis et al., Blood 2022)-can identify a subset of patients who may attain long-term survival without allogeneic hematopoietic stem cell transplantation (allo-HSCT).

The therapeutic strategy consists of a sequential three-phase approach:

Induction: Initial therapy combines the FLT3 inhibitor gilteritinib with venetoclax and azacitidine (the GVA regimen). This synergistic approach targets leukemia through concurrent inhibition of FLT3 and BCL-2 pathways, aiming to achieve high rates of complete remission and deep molecular clearance.

Consolidation: Patients who achieve deep FLT3-ITD negativity, as assessed by the "DeepScan" minimal residual disease (MRD) assay after induction therapy, will proceed to consolidation with high-dose cytarabine (2 g/m² twice daily for 3 days) for three cycles, concurrently with gilteritinib.

Maintenance: Patients maintaining deep FLT3-ITD negativity will receive gilteritinib monotherapy at 120 mg daily for 3 months. Those with detectable mutations will be withdrawn from the study.

A key innovation of this trial is the implementation of "DeepScan," a next-generation sequencing-based assay co-developed with Professor Levis's team. This method detects FLT3-ITD mutations with a sensitivity of up to 10-⁶, surpassing conventional MRD monitoring techniques. It is designed to accurately define a state of deep molecular remission, which serves as the primary biomarker for directing patients toward a transplant-free pathway.

This study challenges the current standard of care, in which allo-HSCT is frequently recommended. By prospectively assessing whether deep molecular responses-induced and maintained through this targeted and chemotherapy-inclusive regimen-can lead to durable survival, the trial aims to provide evidence for a paradigm shift in the treatment of FLT3-ITD-mutated AML, potentially offering a transplant-free alternative for selected patients.

ELIGIBILITY:
Inclusion Criteria:

* Each subject (or their legal representative) must sign an informed consent form (ICF) before any specific study procedures or tests, indicating that he/she understands the purpose and procedures of the study and is willing to participate.
* Age ≥ 18 years or reaching the legal minimum adult age (whichever is greater) and ≤ 60 years (at screening);
* Newly diagnosed acute myeloid leukemia with FLT3-ITD mutation according to the European LeukemiaNet (ELN) 2022 diagnostic criteria (no VAF requirement), with no low-risk or high-risk genetic features as defined by ELN 2022.
* ECOG performance status ≤ 2. Biochemical indicators must be within the following limits within 21 days before randomization and at baseline: ALT and AST ≤ 3× upper limit of normal (ULN); total bilirubin ≤ 3× ULN; serum creatinine ≤ 2× ULN or CrCl ≥ 40 mL/min. LVEF determined by echocardiography is within the normal range (LVEF > 50%).

Exclusion Criteria:

* Diagnosed with acute promyelocytic leukemia (APL), BCR-ABL positive acute myeloid leukemia, or AML secondary to previous chemotherapy or radiotherapy.
* History of other malignancies, except for adequately treated non-malignant skin melanoma, cured in situ tumors, or other solid tumors that have been treated and have had no evidence of disease for at least 2 years.
* Assessed as unfit for intensive chemotherapy based on the following criteria: ECOG performance status ≥ 2 at screening; severe cardiac diseases (e.g., congestive heart failure requiring treatment, ejection fraction ≤ 50%, or chronic stable angina); severe pulmonary diseases (e.g., DLCO ≤ 65% or FEV1 ≤ 65%); creatinine clearance < 45 ml/min (calculated by Cockcroft-Gault equation), liver disease with total bilirubin > 1.5 times the normal upper limit (ULN); any other comorbidities deemed incompatible with intensive chemotherapy by the attending physician.
* Uncontrolled fungal, bacterial, or viral infections.
* Known active clinically relevant liver disease (e.g., active hepatitis B or C); known history of HIV infection (participants should undergo HIV testing before randomization).
* History of allergy to any excipients in gilteritinib tablets.
* Pregnant or breastfeeding women.
* Other conditions deemed unsuitable for this study by the investigator.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite Complete Remission (CRc) Rate after 2 induction cycles | At day 28 of cycle 2 of GVA induction therapy (each cycle is typically 28 days with 2-weeks intervals).
  CRc is defined as the proportion of participants achieving CR or CRi based on 2022 ELN criteria.
  CR: Bone marrow blasts <5%, ANC ≥1.0 x 10⁹/L, platelets ≥100 x 10⁹/L, no extramedullary disease, and transfusion independence.
  CRi: Bone marrow blasts <5%, no extramedullary disease, and insufficient hematologic recovery to qualify for CR.

SECONDARY OUTCOMES:
MRD Negativity Rate | At the time of CRc assessment (at day 28 of cycle 2).
  The proportion of participants who achieve CRc and subsequently achieve Measurable Residual Disease (MRD) negativity, defined as < 0.1% by multiparameter flow cytometry.
Deep Molecular Negativity Rate (for FLT3-ITD) | At the time point for CRc assessment (at day 28 of cycle 2)
  The proportion of participants who achieve deep molecular negative, defined as < 0.0001% (10^-6) via the DeepScan molecular assay, to the patients who achieved CRc
Overall Survival (OS) | follow up 24 months
  Time from enrollment to death from any cause, whichever came first (censored at last follow-up for survivors)
Leukemia-Free Survival (LFS) | follow up 24 months.
  Time from first composed complete remission to relapse or death, whichever occurred first
Molecular Free Survival (mLFS) | follow up 24 months
  The time from first deep molecular negative (FLT3-ITD < 0.0001%) to molecular relapse (above the 0.0001% threshold) or death from any cause
Cumulative Incidence of Relapse (CIR) | follow up 24 months
  The cumulative probability of morphologic relapse, considering death without relapse as a competing risk.
Cumulative Incidence of Molecular Relapse (mCIR) | follow up 24 months
  The cumulative probability of molecular relapse, defined as the re-emergence of FLT3-ITD at or above the 0.0001% threshold, to participants who achieved deep molecular negativity, considering death without molecular relapse as a competing risk.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No